CLINICAL TRIAL: NCT01430481
Title: Comparing Different Preparations and Dosages of Rosehip Powder in Patients With Painful Osteoarthritis of the Knee: An Exploratory Randomised Controlled Trial
Brief Title: Rosehip Powder for Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Frederiksberg University Hospital (Other)
Collaborators: Axellus (Industry); Oak Foundation (Other)
Responsible Party: Principal Investigator, Henning Bliddal, Professor, Frederiksberg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-1-2011-018
Record Dates: First submitted 2011-08-29; First posted 2011-09-08 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Osteoarthritis
Keywords: rosehip; osteoarthritis; pain; knee; RCT
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Rosehip Powder (A) (Active Comparator): 6 capsules of standardized hip powder of Rosa canina made from the seeds and husks of the fruits from a subtype of R. canina hip powder (i.e., rosehip)
  Interventions: Dietary Supplement: Rosehip powder
- New rosehip formulation (B) (Experimental): 6 capsules of modified hip powder of Rosa canina made from the seeds and husks of the fruits from a subtype of R. canina hip powder (i.e., rosehip)
  Interventions: Dietary Supplement: Rosehip powder
- New rosehip formulation in half dose (C) (Experimental): 3 capsules of modified hip powder of Rosa canina made from the seeds and husks of the fruits from a subtype of R. canina hip powder (i.e., rosehip)
  Interventions: Dietary Supplement: Rosehip powder

INTERVENTIONS:
Dietary Supplement: Rosehip powder — The trial is a patient and physician blinded, 12-week, randomized controlled trial (1:1:1). Participants will be randomized into one of 3 groups: 'Standard rosehip powder' (A), 'New rosehip formulation' (B), or 'New rosehip formulation in half dose' (C). Personnel responsible for data collection will be blinded to group assignment. The patients will report on their symptoms every four weeks.
  Other Names: Rosehip; Litomove; Litozin; HybenVital

SUMMARY:
The aim of this study is to compare three combinations of preparations in a comparative trial program on rosehip powder for knee OA. The trial is a comparative, 12-week, randomized, double-blind, active-controlled trial, designed to determine the comparative efficacy and safety of these preparations in patients with pain from knee OA.

DETAILED DESCRIPTION:
Complementary or alternative therapies (incl. nutraceuticals - functional ingredients sold as powders, pills, and other medicinal forms not generally associated with food) for OA are commonly used, and it is therefore important that health care providers are aware of the evidence supporting the claims. One proposed nutraceutical which has shown promising results in OA patients, is the hip powder of Rosa canina.

The findings from a previous meta-analysis of rosehip powder from Rosa canina for symptomatic treatment of OA was a small but potentially relevant reduction of pain and a statistically significant reduction in use of analgesics.

The present study is undertaken to compare two different products, one of which is tested in two different doses, in a non-inferiority design.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age and have clinical evidence (diagnosed according to the American College of Rheumatology [ACR] criteria) and radiographic evidence of OA.
* Eligible patients have a self-reported pain level corresponding to at least 40 mm on a 100 mm VAS when screened

Exclusion Criteria:

* Patients will not be considered eligible if they are considered morbidly obese -having a body mass index (BMI) above 40 kg/m2, concurrent medical or arthritic conditions that could confound evaluation of the index joint, or coexisting disease that could preclude successful completion of the trial.
* Patients who already take a rosehip powder as a dietary supplement; have inability to speak Danish fluently; or have a mental state impeding compliance with the program will not be considered eligible for inclusion.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Pain, Walking on flat surface - range: 0-100 | week 12
  Knee injury and Osteoarthritis Outcome Score (KOOS) subscale item

SECONDARY OUTCOMES:
Pain - range: 0-100 | week 12
  KOOS
Symptoms - range: 0-100 | week 12
  KOOS
Function in daily living - range: 0-100 | week 12
  KOOS
Knee related Quality of life - range: 0-100 | week 12
  KOOS
VAS Pain - 0-100 | week 12
  VAS
VAS Disability - 0-100 | week 12
  VAS
VAS patient global assessment of disease status - 0-100 | week 12
  VAS
VAS physician global assessment of disease status - 0-100 | week 12
  VAS
Physical component summary - range: 0-100 | week 12
  Short-Form-36 score
Mental component summary - range: 0-100 | week 12
  Short-Form-36 score

CONTACTS AND LOCATIONS:
Overall Officials: Henning Bliddal, Professor, Principal Investigator — The Parker Institute, Frederiksberg Hospital, Denmark
Locations (1):
- The Parker Institute, Frederiksberg Hospital, Frederiksberg, Denmark

REFERENCES:
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Background] Christensen R, Bartels EM, Altman RD, Astrup A, Bliddal H. Does the hip powder of Rosa canina (rosehip) reduce pain in osteoarthritis patients?--a meta-analysis of randomized controlled trials. Osteoarthritis Cartilage. 2008 Sep;16(9):965-72. doi: 10.1016/j.joca.2008.03.001. Epub 2008 Apr 14. PMID 18407528
- [Background] Zhang W, Nuki G, Moskowitz RW, Abramson S, Altman RD, Arden NK, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis: part III: Changes in evidence following systematic cumulative update of research published through January 2009. Osteoarthritis Cartilage. 2010 Apr;18(4):476-99. doi: 10.1016/j.joca.2010.01.013. Epub 2010 Feb 11. PMID 20170770
- See also: The Parker Institute, Copenhagen, Denmark — http://www.parkerinst.dk